CLINICAL TRIAL: NCT00532740
Title: A Humanitarian Device Exemption Compassionate Use Protocol of TheraSphere for Treatment of Unresectable Metastatic Cancer to the Liver
Brief Title: Radiolabeled Glass Beads in Treating Patients With Metastatic Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NU 1365-002; P30CA060553 (NIH); NU-1365-002
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: liver metastases; advanced adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All Patients: Patients with metastatic cancer of the liver who are not surgical resection candidates and who will be treated with TheraSphere per institutional standard of care.
  Interventions: Radiation: Yttrium Y 90 glass microspheres

INTERVENTIONS:
Radiation: Yttrium Y 90 glass microspheres — Between 0.2 to 0.5 Curies (200-500-mCi), either single dose to the whole liver, or lobar treatment delivered as a sequence of treatments approximately 30 -90 days apart per treating physician's discretion.

SUMMARY:
RATIONALE: Internal radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Using radiolabeled glass beads to kill tumor cells may be effective treatment for liver cancer that cannot be removed by surgery.

PURPOSE: This phase II trial is studying how well radiolabeled glass beads work in treating patients with metastatic liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide supervised access to treatment with yttrium Y 90 glass microspheres (TheraSphere®) to eligible patients who are not candidates for surgical resection of metastatic intrahepatic carcinoma.
* Evaluate patient experience and toxicities associated with yttrium Y 90 glass microspheres treatment.

OUTLINE: This is a humanitarian device exemption use study.

Patients receive yttrium Y 90 glass microspheres (TheraSphere®) into the liver tumor through a percutaneously placed catheter into the hepatic artery. Patients may receive additional therapy 4-12 weeks after initial treatment at the discretion of the study physician.

After completion of study therapy, patients are followed at 2 weeks, 30 days, and then once a year for approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of metastatic intrahepatic carcinoma

  * Histopathology confirmation may be waived in patients with a radiographically identifiable liver mass AND known laboratory or clinical risk factors for cancer or elevated tumor markers such as AFP
* Unresectable disease
* No portal hypertension with portal venous shunt away from the liver
* FDA approval to receive compassionate use of yttrium Y 90 glass microspheres
* No significant extrahepatic disease representing an imminent life-threatening outcome
* No evidence of potential delivery of > 16.5 mCi (30 Gy absorbed dose) of radiation to the lungs on either of the following:

  * First administration of yttrium Y 90 glass microspheres (TheraSphere ®)
  * Cumulative delivery of radiotherapy to the lungs over multiple treatments

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute granulocyte count ≥ 1,500/µL
* Platelet count ≥ 25,000/μL
* Creatinine ≤ 2.0 mg/dL (unless using non-iodinated contrast or on dialysis)
* Serum bilirubin ≤ 3.0 mg/dL (in some cases where there is an elevated bilirubin, and the tumor may be isolated from a vascular standpoint, treatment may proceed)
* No contraindication to angiography or selective visceral catheterization, including any of the following:

  * History of severe allergy or intolerance to any contrast media, narcotics, sedatives, or atropine, that cannot be controlled using basic angiographic techniques
  * Bleeding diathesis, not correctable by usual forms of therapy
  * Severe peripheral vascular disease that would preclude catheterization
* No severe liver dysfunction or pulmonary insufficiency
* No active uncontrolled infection
* No significant underlying medical or psychiatric illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of any detectable technetium-99 macroaggregated albumin (Tc-99 MAA) flow to the stomach or duodenum after application of established angiographic techniques to stop such flow
* No comorbid disease or condition that would preclude safe delivery of yttrium Y 90 glass microspheres and place patient at undue risk

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* More than 2 weeks since prior surgery
* At least 2 weeks since prior radiosensitizing chemotherapy
* More than 6 weeks since prior carmustine (BCNU) or mitomycin C
* No other concurrent cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic cancer of the liver who are not surgical resection candidates.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2004-12; Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riad Salem, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Rhee TK, Lewandowski RJ, Liu DM, Mulcahy MF, Takahashi G, Hansen PD, Benson AB 3rd, Kennedy AS, Omary RA, Salem R. 90Y Radioembolization for metastatic neuroendocrine liver tumors: preliminary results from a multi-institutional experience. Ann Surg. 2008 Jun;247(6):1029-35. doi: 10.1097/SLA.0b013e3181728a45. PMID 18520231
- [Result] Sato KT, Lewandowski RJ, Mulcahy MF, Atassi B, Ryu RK, Gates VL, Nemcek AA Jr, Barakat O, Benson A 3rd, Mandal R, Talamonti M, Wong CY, Miller FH, Newman SB, Shaw JM, Thurston KG, Omary RA, Salem R. Unresectable chemorefractory liver metastases: radioembolization with 90Y microspheres--safety, efficacy, and survival. Radiology. 2008 May;247(2):507-15. doi: 10.1148/radiol.2472062029. Epub 2008 Mar 18. PMID 18349311